CLINICAL TRIAL: NCT02125422
Title: Neurophysiological Study of tDCS Effects in Healthy Volunteers
Acronym: tDCSHV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CB-1200
Record Dates: First submitted 2014-04-18; First posted 2014-04-29 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cefaly tDCS (Experimental): Cathodal Cefaly tDCS is delivered over the visual cortex at 2 mA of intensity, for 20 minutes, for 5 consecutive days in 9 HV. The anode is placed over the left DLPFC.
  2 mA anodal tDCS is delivered over the visual cortex, for 20 minutes, for 5 consecutive days in 9 HV
  Interventions: Device: Cefaly tDCS

INTERVENTIONS:
Device: Cefaly tDCS — Cefaly tDCS (transcranial direct current stimulation) is able to modify cortical excitability, in particular anodal tDCS increases it. The side effects of tDCS are minor, especially sensations of itching and scalp paresthesias.

SUMMARY:
Transcranial direct current stimulation is a tool to modulate cortical excitability.

DETAILED DESCRIPTION:
Anodal transcranial direct currenti stimulation over visual cortex is able to decrease the thermo-nociceptive sensibility and thermonociceptive potentials, whilst cathodal transcranial direct current stimulation has the opposite effect, it decreases VEP amplitude and habituation. This neuromodulation technique is probably a tool in the prevention in episodic and chronic migraine.

The aim of the study is to study short and long term effect of tDCS over pain treshold, contact heat evoked potentials, blink reflex and visual evoked potentials in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* age below 18 or above 65 years
* personal history of recurrent headache or other neurological diseases especially seizures,
* familial history of recurrent headache
* child migraine equivalents (motion sickness, cyclic vomiting or recurrent abdominal pain, somnambulism etc.. . .)
* chronic pain syndromes
* analgesics intake at the time of recording
* contra-indications to tDCS neurostimulation (metal prosthetics in the head or internal stimulation like a pacemaker).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Neurophysiological mesures changes | up to 1 month
  Modifications in neurophysiological test after direct current stimulation

OTHER OUTCOMES:
VEP changes | up to 1 month
  Evaluation of changes in latency, amplitude, slope and habituation
Blink changes | up to 1 month
  Evaluation of changes in latency, amplitude, slope and habituation
CHEPS changes | up to 1 month
  Evaluation of changes in latency, amplitude, slope and habituation
Quantitave Sensory Testing | up to 1 month
  Evaluation of changes in thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Magis, MD, Principal Investigator — University of Liege; Jean Schoenen, MD, Principal Investigator — University of Liege
Locations (1):
- Roberta Baschi, Liége, Liége, Belgium